CLINICAL TRIAL: NCT00910377
Title: Effect of Intervention About Breastfeeding and Complementary Feeding in Adolescent Mothers and Their Grandmothers
Brief Title: Adolescent Mothers, Grandmothers, Breastfeeding and Complementary Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Elsa Regina Justo Giugliani, MD, PhD, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-389
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Breastfeeding; Weaning
Keywords: breastfeeding; exclusive breastfeeding; lactation counseling; teenagers; complementary food; adolescent; caregivers
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- visit with grandmother (Experimental): Teenagers mothers and their grandmothers receive counseling sessions about breastfeeding and complementary feeding.
  Interventions: Behavioral: counseling sessions
- visit without grandmother (Experimental): Teenagers mothers don´t live with their grandmothers and receive counseling sessions about breastfeeding and complementary feeding.
  Interventions: Behavioral: counseling sessions
- no visit with grandmother (No Intervention): Teenagers mothers live with their grandmothers and don´t receive counseling sessions about breastfeeding and complementary feeding.
- no visit without grandmother (No Intervention): Teenagers mothers don´t live with their grandmothers and don´t receive counseling sessions about breastfeeding and complementary feeding.

INTERVENTIONS:
Behavioral: counseling sessions — The intervention groups received counseling sessions about breastfeeding and complementary feeding at maternity ward and at home with 7,15,30,60 and 120 days.
  Other Names: Group one- no grandmother and no intervention; Group two- no gradmother and with intervention; Group three - with grandmother and no intervention; Group four- with grandmother and with intervention
  Arms: visit with grandmother; visit without grandmother

SUMMARY:
The purpose of this study is to determine whether counseling sessions on breastfeeding for adolescent mothers and their grandmothers in the maternity ward and at home are effective in to improve the exclusive and total breastfeeding rates during the first six month, as well as the convenient timing of supplementary feeding introduction.

DETAILED DESCRIPTION:
Despite the recognized value of exclusive breastfeeding during the first months of a child's life and efforts for promoting this practice, rates for this pattern of breastfeeding in Brazil are below those recommended by the World Health Organization(WHO), which advocates exclusive breastfeeding during the first 6 months. The last national survey about the prevalence of breastfeeding revealed a median duration of 10 months. However , the length of exclusive breastfeeding was only 23 days.

A lot of studies identified maternal age as predictor of breastfeeding. In African, Asian, Latin American and the Pacific societies, older women, or grandmothers,traditionally have considerable influence on decisions related to maternal and child health at the household level.

Considering all that, interventions intended to increase frequency of breastfeeding, particularly exclusive breastfeeding. However, there are few studies on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent mothers
* Mothers living in the city of Porto Alegre
* Healthy nontwin newborns with birth weight equal or greater than 2500g

Exclusion Criteria:

* Mothers living with mother-in-law
* Mother-infant pairs that were unable to stay together due to a health concern in either the mother or infant
* Mammaplasty reductive

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 344 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of exclusive and total breastfeeding | First year

SECONDARY OUTCOMES:
Pattern of complementary feeding | one year

CONTACTS AND LOCATIONS:
Overall Officials: ELSA REGINA J GIUGLIANI, MD,PhD,IBCLC, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] da Silva CF, Nunes LM, Schwartz R, Giugliani ER. Effect of a pro-breastfeeding intervention on the maintenance of breastfeeding for 2 years or more: randomized clinical trial with adolescent mothers and grandmothers. BMC Pregnancy Childbirth. 2016 May 3;16:97. doi: 10.1186/s12884-016-0878-z. PMID 27141951
- [Derived] Schwartz R, Vigo A, de Oliveira LD, Justo Giugliani ER. The Effect of a Pro-Breastfeeding and Healthy Complementary Feeding Intervention Targeting Adolescent Mothers and Grandmothers on Growth and Prevalence of Overweight of Preschool Children. PLoS One. 2015 Jul 10;10(7):e0131884. doi: 10.1371/journal.pone.0131884. eCollection 2015. PMID 26161657
- [Derived] Dias de Oliveira L, Justo Giugliani ER, Cordova do Espirito Santo L, Meirelles Nunes L. Counselling sessions increased duration of exclusive breastfeeding: a randomized clinical trial with adolescent mothers and grandmothers. Nutr J. 2014 Jul 17;13:73. doi: 10.1186/1475-2891-13-73. PMID 25033743
- [Derived] de Oliveira LD, Giugliani ER, Santo LC, Nunes LM. Impact of a strategy to prevent the introduction of non-breast milk and complementary foods during the first 6 months of life: a randomized clinical trial with adolescent mothers and grandmothers. Early Hum Dev. 2012 Jun;88(6):357-61. doi: 10.1016/j.earlhumdev.2011.09.010. Epub 2011 Oct 15. PMID 22001312